CLINICAL TRIAL: NCT06319326
Title: Intestinal Perfusion After Feeding in Preterm and Term Infants
Status: Not yet recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Xiamen Children's Hospital (Other)
Responsible Party: Principal Investigator, Agostino Pierro, Dr, The Hospital for Sick Children
Other Study IDs: Postfeed Intestinal Perfusion
Record Dates: First submitted 2024-02-22; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Premature; Necrotizing Enterocolitis
Keywords: intestinal perfusion; postprandial intestinal perfusion; Color Doppler abdominal ultrasound
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing | interventions — Postprandial Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm infants: Preterm infants (≤33 weeks gestational age) of any birth weight receiving full bolus enteral feeding, aged 1-4 weeks.
  Interventions: Other: Evaluation of intestinal perfusion with color Doppler abdominal ultrasound before and after feeding.
- Term infants: Term infants of any birth weight aged 1-4 weeks.
  Interventions: Other: Evaluation of intestinal perfusion with color Doppler abdominal ultrasound before and after feeding.

INTERVENTIONS:
Other: Evaluation of intestinal perfusion with color Doppler abdominal ultrasound before and after feeding. — This is an observation study involving measurement of intestinal perfusion with color Doppler abdominal ultrasound before and after feeding. No intervention is given to study participants.
  Other Names: No intervention.

SUMMARY:
This is a pilot exploratory observational prospective cohort phase I study. In this study, we will gather preliminary data to evaluate (i) the magnitude of changes in blood flow in the bowel before and after feeding and (ii) the differences between preterm and term infants.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is the most devastating intestinal disease which remains a major unsolved clinical challenge in neonatology. NEC is predominantly a disease of preterm or extremely preterm infants. NEC results in high mortality, neurodevelopmental impairment, intestinal failure, and reduced quality of life.

Prematurity and enteral feeding are two of the most important risk factors for NEC. More than 90% of infants with NEC have been enterally fed, suggesting that feeding is an important priming step in making the intestine vulnerable to NEC. Absorption of nutrients is energy-consuming and results in an increased oxygen demand after feeding, followed by an increase in intestinal blood flow above baseline (known as postprandial hyperemia). Our preclinical studies have shown an intriguing discovery, that prematurity is associated with a remarkably reduced intestinal response to feeding, which predisposes the intestine to NEC.

However, there is lack of reliable clinical evidence to compare the magnitude of difference in postprandial intestinal blood flow in human preterm versus term infants. If preterm infants do in fact demonstrate a diminished intestinal blood flow response to feeding, this will shed light on the need for interventions in the feeding protocol of this vulnerable population to prevent the development of NEC.

This study is a phase I exploratory prospective cohort study. We will gather preliminary data to evaluate (i) the magnitude of changes in blood flow in the bowel before and after feeding and (ii) the differences between preterm and term infants.

In a cohort of 20 patients (10 preterm, 10 term), we will evaluate feeding-related perfusion of the superior mesenteric artery and bowel wall immediately before and 60-minutes after feeding.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (≤33 weeks gestational age) of any birth weight receiving full bolus enteral feeding.

Exclusion Criteria:

* Neonates receiving bolus enteral feeds lasting >30 minutes or continuous enteral feeds will be excluded to avoid overlapping or close timing between pre- and post-prandial intestinal perfusion measurements.
* Large patent ductus arteriosus (PDA)
* Major congenital malformations
* Suspected genetic syndrome
* Ssuspected or confirmed infection
* Fraction of inspired oxygen of ≥0.60 at enrollment
* Confirmed diagnosis of necrotizing enterocolitis diagnosis. NEC will be diagnosed when at least two of the following clinical signs and one radiological sign will be present: (i) Clinical signs (1. abdominal distension; 2. abdominal tenderness; 3. abdominal discoloration; 4. blood in stool). (ii) Radiological signs (1. Pneumoperitoneum; 2. pneumatosis; 3. portal venous gas).

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consists of 2 cohorts:
  * Preterm infants (≤33 weeks gestational age at birth) of any birth weight receiving full bolus enteral feeding.
  * Term infants of any birth weight aged 1-4 weeks.
  The sources of preterm infants are level III/IV neonatal intensive care units at Xiamen Children's Hospital and the Hospital for Sick Children. The source of the cohort of term infants will be Level II neonatal ward at Children's Hospital of Fudan University (Xiamen Branch), Xiamen Children's Hospital and the Hospital for Sick Children.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-02 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Time-averaged mean velocity of the superior mesenteric artery | Measured immediately before and 60 minutes after feeding
  Abdominal ultrasound is used to measure the percent change in time-averaged mean velocity (TAMV) of the superior mesenteric artery (SMA) between pre and post-prandial assessments.

SECONDARY OUTCOMES:
Bowel wall perfusion | Measured immediately before and 60 minutes after feeding
  Color Doppler abdominal ultrasound is used to measure changes in peripheral perfusion of the bowel wall pre- and post-prandially.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University (Xiamen Branch), Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Y, Koike Y, Chi L, Ahmed A, Miyake H, Li B, Lee C, Delgado-Olguin P, Pierro A. Formula feeding and immature gut microcirculation promote intestinal hypoxia, leading to necrotizing enterocolitis. Dis Model Mech. 2019 Dec 9;12(12):dmm040998. doi: 10.1242/dmm.040998. PMID 31704804
- [Background] Chen Y, Koike Y, Miyake H, Li B, Lee C, Hock A, Zani A, Pierro A. Formula feeding and systemic hypoxia synergistically induce intestinal hypoxia in experimental necrotizing enterocolitis. Pediatr Surg Int. 2016 Dec;32(12):1115-1119. doi: 10.1007/s00383-016-3997-8. Epub 2016 Nov 4. PMID 27815640